CLINICAL TRIAL: NCT03777449
Title: The Morphology of the Peri-Implantitis Defects: A Cone-Beam Computed
Brief Title: The Morphology of the Peri-Implantitis Defects: A Cone-Beam Computed Analysis
Status: Completed | Type: Observational
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Other Study IDs: 18002909-12/2018
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vertical bone loss: Infra-osseous defects
  Interventions: Radiation: CBCT
- Horizontal bone loss: Supra-osseous defects
  Interventions: Radiation: CBCT
- Combined bone loss: Combined supra-osseous and infra-osseous defects

INTERVENTIONS:
Radiation: CBCT — Patients will be taken a CBCT as a diagnostic tool to monitor peri-implant bone loss. This is a tool used on the daily basis for the evaluation of peri-implant bone loss. Patient will not be exposed to further radiation but the regular one.
  Groups: Horizontal bone loss; Vertical bone loss

SUMMARY:
To study the morphology of the peri-implant defects using cone-beam computed tomography based on a priori case definition of peri-implantitis (≥3mm of radiographic bone loss + inflammatory clinical parameters)

Diagnosis of peri-implantitis requires:

* Presence of bleeding and/or suppuration on gentle probing.
* Increased probing depth compared to previous examinations.
* Presence of bone loss beyond crestal bone level changes resulting from initial bone remodeling.

In the absence of previous examination data diagnosis of peri-implantitis can be based on the combination of:

* Presence of bleeding and/or suppuration on gentle probing.
* Probing depths of ≥6 mm.
* Bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant.

DETAILED DESCRIPTION:
Nowadays, several radiographic techniques are available to investigate the peri-implant bone morphology by two-dimensional radiographs such as panoramic radiography and intraoral radiography, or three-dimensional techniques such as computer tomography and cone beam computer tomography (CBCT) (Harris et al. 2012). CBCT provides high-contrast 3D visualization of bone beds; however, artifacts caused by the metallic character of implants could disguise information around implants. The diagnostic outcomes of CBCT imaging of peri-implant bone loss have been related to the type of study and defect morphology (Pelekos et al., 2018). The ex vivo studies (cadaver models), considering sensitivity and specificity reported good values for both circumferential and infrabony defects but lower for dehiscences (de-Azevedo-Vaz et al., 2013, Kamburoglu et al., 2013). Contrastingly, CBCT imaging for defect analysis in animal studies showed positive correlation with histology but tend to overestimate (Fienitz et al., 2012, Golubovic et al., 2012) or underestimate (Corpas Ldos et al., 2011, Ritter et al., 2014) the size of the defect. This variability in the measurement is mainly dependent on the different configuration, location or size of the defect. and also by the scattering, beam hardening artifacts, energy settings, exposure time, field of view.

Hence, it is aimed at assessing the morphology of the peri-implant defects using CBCT

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 80 years of age
* Partial/complete edentulism missing one or more teeth and having it restored with implant-supported prosthesis
* No antibiotic in the last 2 months previous to examination
* >3 year after prosthesis delivery

Exclusion Criteria:

* Uncontrolled systemic disease
* Cemented-retained restorations
* Patients with uncontrolled/active periodontal disease in need of periodontal treatment
* Pregnant patients
* Zygomatic implants
* Implants placed in regenerated/augmented bone
* Patients taking medications known to modify bone metabolism or known to have degenerative diseases of bone (hyperparathyroidism, osteoporosis), vitamin D, patients who had taken antibiotics, NSAIDS or corticosteroids for more than two weeks in the past 3 months before examination

Age Groups: Child, Adult, Older Adult
Study Population: Healthy partially/complete edentulous having previously received screw-retained implants for oral rehabilitation for ≥3 years.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Morphology | 6 months
  Morphology of the peri-implant defects ivy number of existing bone walls present (1, 2, 3 or 4)

SECONDARY OUTCOMES:
Severity of the peri-implant bone loss | 6 months
  Distance in mm from the top of the implant down to the defect base

CONTACTS AND LOCATIONS:
Locations (1):
- CICOM, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Monje A, Pons R, Insua A, Nart J, Wang HL, Schwarz F. Morphology and severity of peri-implantitis bone defects. Clin Implant Dent Relat Res. 2019 Aug;21(4):635-643. doi: 10.1111/cid.12791. Epub 2019 May 14. PMID 31087457